CLINICAL TRIAL: NCT06497426
Title: Efficacy of a Water Intervention in the Improvement of Anabolic Resistance and Some Physiologic Adaptive Water Conservation Mechanisms in Institutionalized Aged Population. A Randomized Controlled Trial.
Brief Title: Efficacy of a Water Intervention in Institutionalized Aged Population.
Acronym: FIS22-AC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14/23
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water intake intervention (Experimental): During one week, participants will be asked to drink 30 (for women) or 35 (for men) ml of water/Kg of weight/day distributed homogeneously during the day. The water requirements of subjects with overweight will be calculated with the corrected weight using the Wilkens formula. Water will be provided in the form of 1L bottles and recommendations about the amount of water to intake will be individualized and indicated by a mark on the bottle. Water intake will be supervised by a nurse/nurse assistant/dietitian team to ensure adherence, and registered to assess intervention compliance. This water intake will be apart from usual meals. A dietitian will prepare the daily amount of mineral water in 1 liter bottles to facilitate the intervention supervision and compliance. All bottles will be identified by NID and date and will be retired and replaced every day at 8-9 am for compliance assessment. Participants will be asked to drink only the provided water.
  Interventions: Other: Study intervention
- Control intervention (No Intervention): Usual clinical practice with no especial attention to hydration. Participants will be able to freely drink whatever they want (ad libitum). Participants in the control group will be provided with 2 bottles of 1L (2L of water) every day, and more water will be provided if requested. Daily water intake will also be quantified.

INTERVENTIONS:
Other: Study intervention — Participants will be asked to drink water. Water intake will be supervised by a nurse/nurse assistant/dietitian team to ensure adherence, and registered to assess intervention compliance.
  Arms: Water intake intervention

SUMMARY:
Background: As a person ages, there is a decrease in the body's ability to respond to feeding and exercise anabolic stimuli and to produce muscle proteins. Causes of this anabolic resistance in aged population are not well known. Total body water also decreases with age and has been related with muscle mass, strength and performance.

Objective: The aim of this study is to assess the effect of a water intervention on anabolic resistance and on some physiological adaptive response to water loss indicators in institutionalized aged population. Methodology: Design and population: randomized controlled trial with two parallel arms in ≥65-year-old institutionalized subjects. Study intervention: supervised water ingestion (30-35 ml/kg/day) during 7 consecutive days. Control intervention: usual care (water ingestion ad libitum). Main outcome measures: a)anabolic resistance (nitrogen balance, 3-methyl-histindine, urea excretion, plasmatic and urinary urea and urea/high index), b) indicators of physiological adaptive mechanism to water conservation (copeptin, sympathetic tone, inflammatory indicators, anabalic and catabolic hormones), c)muscle mass (according to bioimpedance analysis), grip strength (JAMAR dynamometer), sarcopenia (according to EWGSOP 2 criteria), and d) clinical recovery.

Controls and follow-up: at 1 week and hospital discharge.

DETAILED DESCRIPTION:
Population ageing, frailty and sarcopenia:

Population aging is one of the main challenges faced by Western societies. The lengthening of life expectancy has led to an increase in the need for medical and social care. Frailty is one of the most relevant consequences of the population ageing. Frailty is a well established geriatric syndrome characterized by a decrease in the body's reserves and its ability to respond against external stressors. It results in a decline in the function of several organs and systems that leads to greater vulnerability to suffer diseases, adverse health outcomes, functional decline, falls, disability or dependency. Frail subjects are in an increased risk of hospitalization, nursing home admission and mortality. Prevalence of frailty increases with age and can reach 50% in the population over 80 years old. Frailty evolves but is also potentially reversible (and treatable), especially in its initial stages. For all these reasons, frailty is considered today a real public health problem and a social threat that needs urgent attention. However, the ultimate causes of frailty is still unknown. Frailty is related with reduced muscle mass and function and with sarcopenia, which is defined as the loss of muscle function (strength or performance) accompanied by loss of muscle quantity or quality (EWGSOP2). Sarcopenia is a main determinant of functional decline, disability and dependency in aged population. Functional dependency has a prevalence of 20% in ≥65 year old population and of 30% in ≥75 years old population, with clear predominance in women. Different related factors contribute to sarcopenia, including changes in protein kinetics, hormonal regulation, grow factors, vascularization, inflammation, mitochondrial function, nutrition or physical exercise, but its pathophysiology is not completely understood. Currently, there is no effective drug to treat sarcopenia, but resistance exercises and nutritional measures are effective anabolic stimuli to maintain or ameliorate muscle function.

Dehydration in aged population:

Water is a main component in the human body and an essential nutrient for life and health. Water represents approximately 50-60% of total body weight in adults and has fundamental structural, metabolic, transport and thermo regulation functions. Water in the body is distributed in the extracellular and intracellular compartments and flows from one compartment to the other through a group of transmembrane proteins called aquaporines (AQP) by diffusion process guided by osmotic pressure. Water balance in human body is tightly regulated by the kidneys, which can concentrate or dilute urine depending on the metabolic waste and water intake. Water losses occur mainly in urine and sweat, but also through feces and breathing. Vasopressin (AVP) plays a fundamental role in water homeostasis by, in response to osmotic and pressure stimuli, increasing renal water reabsorption. From adulthood, there is a progressive decline in the water content of the body. Muscle is the main water reservoir in the organism. Loss of muscle mass is related with loss of total body water, especially when there is an increase in fat mass. Nonetheless, there are reasonable doubts about whether loss of muscle mass is responsible for loss of body 5 water or, by contrary, loss of body water is responsible for loss of muscle mass. Causes of the progressive chronic dehydration process in aged population are not well known, but may include a decreased water intake, decreased water absorption, decreased capacity to concentrate urine because of peripheral resistance to AVP or increased water losses due to medications or other circumstances such as situations of high heat or physical exercise. The renal solutes load (RSL) is the amount of metabolic waste by-products that must be eliminated by the kidney, while the obligatory urine water volume (OUV) is the minimum amount of water eliminated by the kidneys that is required to eliminate the RSL. OUV depends on the RSL and the renal capacity to concentrate urine. If the ability to concentrate urine is reduced, then the amount of urine should be increased to ensure elimination of waste products, but water intake should also be increased to avoid dehydration. It is difficult for aged population to increase water intake (because of anorexia, decreased thirst, urine incontinence, prostatic symptoms, etc.) so they are at increased risk of dehydration. Prevalence of dehydration in the elderly is usually under-recognised and has been estimated at 20%- 30% and is associated with greater disability, morbidity and mortality. There are no clear and objective clinical signs of early dehydration in the elderly, but plasma and urinary osmolaritiescan be considered the gold standard for a diagnosis of dehydration. In a population-based observational study (PI19/00500) with 237 subjects aged 70 years or over our group showed that: a) urine osmolarity was lower in women and decreases with age; b) plasma hyperosmolarity (>295 mOsm/L) was present in no women but in 4.5% of men, and was significantly 14 times greater in the older group; c) prevalence of resistance to AVP was 12.3%, 10.4% in subjects aged 70-79 vs 20.7% in subjects aged ≥80; and d) subjects with resistance to AVP presented higher plasma osmolarity and a prevalence of plasma hyperosmolarity of 10.0% (compared to 0.7%; p=0.004, in subjects with no resistance to AVP). Thus, the investigators concluded that urine concentration capacity decreases and plasma hyperosmolarity increases after the age of 80 years, and that peripheral resistance to AVP, with an overall prevalence of 12.3% in ≥70 years old population, greatly increases the risk of plasma hyperosmolarity (intracellular dehydration). Dehydration represents a heterogeneous group of conditions and its assessment is a major clinical challenge due to a complex, varying pathophysiology, non-specific clinical presentations and the lack of international consensus on its definition and diagnosis. Dehydration should mainly refer to hypertonic or isotonic dehydration. Hypertonic dehydration is due to a pure water deficit (without deficit of solutes) because insufficient dinking, excessive sweating or inability to concentrate urine (typical in aged population). It results in an increase in plasmatic osmolarity and a movement of water from intracellular to extracellular spaces (fluid loss is primarily from within cell). In contrast, isotonic dehydration with water and solute loss due to acute blood loss, vomiting or secretory diarrhea and no osmotic gradient between fluid compartments, is characterized by extracellular volume loss and intravascular fluid depletion (hipovolemia), which requires volume resuscitation with salt-containing fluid.

Hyperosmotic stress and its consequences:

Extracellular (plasmatic) osmolarity should be kept between 285-295 mOsm/L to be compatible with life. The increase in extracellular osmolarity has important harmful effects as favors intracellular dehydration (cellular contraction), which affects the 6 structure and function of proteins and alters intracellular enzymatic activity. Cell damage is proportional to osmotic imbalance and may lead to cell death. Osmotic balance is regulated primarily by the AVP, which stimulates renal water reabsorption and urinary concentration. However, as mentioned before, aged population has reduced capacity to concentrate urine and exhibit some peripheral resistance to AVP. Cells have developed other mechanisms to compensate extracellular hyperosmolarity and restore osmotic equilibrium such as the activation of ion transporters, the synthesis of osmolytes (mainly urea), the induction of gene expression of AQP, rearrangement of the cytoskeleton, or the activation of antioxidant enzymes. Moreover, increased extracellular osmolarity (or hyperosmotic stress) has been related with inflammation, diabetes, insulin resistance and metabolic disorders, chronic kidney disease and nephrolithiasis, cardiovascular diseases and oxidative stress, all of them also related with frailty. However, the effect of hyperosmotic stress and cell dehydration on muscle has been poorly studied in aged population.

Adaptive response to dehydration:

Some evidences suggest that the inability to concentrate urine induce an extrarenal compensatory response to prevent dehydration. Chronic water loses led to an increase in plasma osmolality, mainly explained by an increase in plasma urea concentration. An experiment in 5/6 Nx rats with renal mass ablation showed diminished capacity to concentrate urine, increased urine volume, increased plasma urea concentration and in the absence of reduced renal urea excretion. These results suggest that renal fluid loss had triggered a compensatory hepatic response with urea osmolyte production in an effort to stabilize body water content. These rats with renal water loss increased transfer of nitrogen into the urea cycle mainly by the catabolism of the aminoacids arginine and BCAAs and the dipeptides anserine and carnosine. They explote their muscle and muscle energy and nitrogen reservoirs to support hepatic urea osmolyte production in an attempt to retain water. Moreover, this study shows an increased peripheral vascular resistance due to an increased generation of endothelial nitric oxide (NO) synthase inhibitors (which increases the vascular tone), oxidative stress, an increase in plasma AVP levels and increased norepinephrine excretion (indicating increased sympathetic tone). Physiological adaptation to renal water loss in 5/6 Nx rats also included cutaneous vasoconstriction in an effort to reduce trans epithelial water loss, but at expenses of elevated blood pressure.

Anabolic resistance:

Maintenance of skeletal muscle mass depends on a balance between muscle protein synthesis (MPS) and muscle protein breakdown (MPB). Age and catabolic pathologies result in loss of muscle mass because a negative imbalance in protein turnover (low MPS or high MPB). Anabolic resistance, that is, loss of sensitivity to main anabolic stimuli, such as feeding or exercise, may be responsible for the age-related decline in MPS. In healthy muscle, protein consumption stimulates MPS in a dose-response manner, with excess dietary amino acids being catabolized. The MPS response to protein intake is enhanced with resistance 7 exercise performed before ingestion. The aminoacid composition of ingested protein is also an anabolic stimulus for MPS, with branched-chain amino acids (BCAAs) content (leucine, isoleucine and valine) being an especially potent stimulator of postprandial MPS. The anabolic response to exercise and feeding is observed within several hours after acute stimulus and is mediated by insulin, IGF-1 and BCAAs, and regulated by the mammalian/mechanistic target of rapamycin (mTOR). In contrast, MPB seems to be less sensitive to dietary aminoacid availability. There is a decreased MPS response to protein ingestion in older adults but its causes are not well established. A reduction of approximately 10% in dietary protein absorption has also been observed in aged adults, so increase protein ingestion to 1.2g/kg/day is recommended in this population. Moreover, distributing protein ingestion throughout the day, ingesting quality proteins and exercise, especially resistance exercise, prior protein ingestion have shown to improve sensitivity to MPS. It is imperative for older adults to exercise and adhere to healthy eating patterns to prevent anabolic resistance, loss of muscle mass and sarcopenia, but these recommendations are difficult for most aged people to adhere or comply with.

On the other hand, regardless of age, obesity, cancer and other inflammatory diseases can also reduce the MPS response to anabolic stimuli.

Study justification:

Muscle mass starts to decline around the age of 40 and this loss increases progressively with age. The loss of muscle mass involves both a reduction in the number of muscle fibers and a decrease in their size, causing atrophy and being responsible for sarcopenia and functional decline. As a person ages, certain changes take place in the body that play a role in the development of sarcopenia. One of these changes is a decrease in the body's ability to respond to feeding and exercise anabolic stimuli and to produce muscle proteins, which has been called anabolic resistance. Causes of anabolic resistance in aged population are not well known. Inflammation or age-related anabolic hormone decline may be responsible for a decrease in muscle mass. It is known that levels of testosterone, GH, insulin-like growth factor (IGF-1) or insulin may decrease with age and affect muscle growth and mass. Other age-related factors that can contribute to sarcopenia are the behavior ones, such as a sedentary lifestyle and poor dietary habits with poor protein ingestion.

Moreover, as the age increases, the amount of total body water decreases, and older people have a higher risk of dehydration due to lower water intake and increased water loses. Muscle is a main reservoir of water in the body and, therefore, it is logical that a decrease in muscle mass is accompanied by decrease in total body water. However, it is unclear whether water loss is the consequence or is the cause of the loss of muscle mass and function. Numerous studies have shown that even small losses of body water can negatively affect muscle strength, endurance, and maximal oxygen uptake. The investigatorshypothesize that dehydration, specifically intracellular dehydration due to hyperosmotic stress caused by higher loss of water than solutes (typical of aging), may be related to anabolic resistance, decreased protein synthesis and sarcopenia. The physiological response to increased plasma osmolarity includes, in addition to an inflammatory response, the synthesis of urea osmolyte to further increase plasma osmolarity in an attempt to retain water. This urea synthesis consumes energy and nitrogen from amino acids, has catabolic effects 8 and contributes to anabolic resistance. The investigatorshypothesize that AVP resistance and the loss in the ability to concentrate urine is responsible for hyperosmotic stress in aged population, that dehydration and high plasmatic osmolarity is responsible for anabolic resistance, and that anabolic resistance is responsible for sarcopenia, frailty and functional decline in aged population. If dehydration causes anabolic resistance,

ELIGIBILITY:
Inclusion Criteria:

* subjects ≥65 years,
* institutionalized in a nursing home or in a convalescence unit in a socio sanitary center,
* who give their informed consent.

Exclusion Criteria:

* acute infectious disease,
* exacerbation of a chronic inflammatory disease
* less than 3 weeks from surgery,
* hepatic cirrhosis,
* chronic renal failure (with glomerular filtrate <40),
* decompensate heart failure with edema in lower-limbs or acute pulmonary edema,
* active neoplasia,
* in palliative care or life expectancy less than 6 months,
* advanced dementia (GDS>5),
* dysphagia,
* carrier of bilateral hip or knee prostheses, heart pacemaker
* serum therapy,
* Users of parenteral nutrition or nasogastric tube nutrition, and
* users of diapers (if they are not regular urinary tract carriers).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Nitrogen balance | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Nitrogen balance (NB) measures the difference between nitrogen intake and the amount excreted in feces, urine, and sweat. Losing 13 more nitrogen than we consume in the diet would result in a negative NB. This situation indicates that the body is losing protein and does not have the adequate amount of nitrogen to build and repair cells and tissues.
Plasmatic and urinary urea concentration | Baseline, 1 week of follow-up, 2 weeks of follow-up
  an increase of both may suggest dehydration when there is no antecedent of renal failure
Urea | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Fractional excretion of urea
Creatinine-height index | Baseline, 1 week of follow-up, 2 weeks of follow-up
  The creatinine-height index determines the relationship between the observed and expected creatinine clearance for an adult of the same age and height.

SECONDARY OUTCOMES:
Inflammatory parameters | Baseline, 1 week of follow-up, 2 weeks of follow-up
  plasmatic CRP and IL-6 levels
Sympathetic tone | Baseline, 1 week of follow-up, 2 weeks of follow-up
  plasmatic norepinephrine levels
Plasma copeptin levels | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Copeptin, a 39-amino acid-long peptide derived from the c-terminus of pre-pro-hormone of AVP, neurophysin II, and copeptin, is co-released with AVP from the hypothalamus and is considered a reliable AVP surrogate
Plasmatic anabolic hormones | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Testosterone, GH, IGF-1, Insulin
Plasmatic catabolic hormones | Baseline, 1 week of follow-up, 2 weeks of follow-up
  cortisol, ACTH
Plasmatic osmolarity | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Plasmatic osmolarity
Urinary osmolarity | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Urinary osmolarity
BIA hydration parameters | Baseline, 1 week of follow-up, 2 weeks of follow-up
  Total body water, extracellular water (ECW) and intracellular water (ICW)

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No